CLINICAL TRIAL: NCT00000466
Title: Postmenopausal Estrogen/Progestin Interventions (PEPI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: National Institute on Aging (NIA) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 55; U01HL040232 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-07

CONDITIONS: Bone Diseases; Cardiovascular Diseases; Coronary Disease; Diabetes Mellitus; Heart Diseases; Hypercholesterolemia; Hypertension; Myocardial Ischemia; Osteoporosis; Thrombosis; Postmenopause
MeSH Terms: conditions — Bone Diseases; Cardiovascular Diseases; Coronary Disease; Diabetes Mellitus; Heart Diseases; Hypercholesterolemia; Hypertension; Myocardial Ischemia; Osteoporosis; Thrombosis | interventions — Estrogens, Conjugated (USP); Medroxyprogesterone; Progesterone; Estrogen Replacement Therapy

INTERVENTIONS:
Drug: estrogens, conjugated
Drug: medroxyprogesterone
Drug: progesterone
Drug: estrogen replacement therapy

SUMMARY:
To assess the effects of various postmenopausal estrogen replacement therapies on selected cardiovascular risk factors, including high density lipoprotein cholesterol, systolic blood pressure, fibrinogen, and insulin and on osteoporosis risk factors. Conducted in collaboration with the National Institute of Child Health and Human Development, the National Institute of Arthritis and Musculoskeletal and Skin Diseases, The National Institute of Diabetes and Digestive and Kidney Diseases, and the National Institute on Aging. The extended follow-up is for 3 years focusing on endometrium and breast evaluation.

DETAILED DESCRIPTION:
BACKGROUND:

The life expectancy of American women is 78 years. More than one-third of those years are postmenopausal, during which time the risk of coronary heart disease is increased. The current United States estimate of more than 40 million women over the age of 50 indicates a large segment of the population at increased risk for coronary heart disease. Heart disease accounts for a third of all deaths in 50-69 year old women. In 1978, for example, approximately 66,000 of the 210,000 deaths in women 50-69 were attributed to heart disease.

Premenopausal women have a lower rate of ischemic heart disease compared to men of similar age. Surgically induced or natural early menopause increases the risk of ischemic heart disease. These facts have focused interest on estrogens as possible mediators of the beneficial effects, and pointed to the need for further study of their relationship to atherosclerosis risk factors.

Estimates from the Lipid Research Clinics Program indicate estrogen use in approximately one third of postmenopausal women. Analysis of Lipid Research Clinics data confirmed that administration of estrogens results in lower plasma low density lipoprotein levels and elevated plasma high density lipoprotein levels. Thus, the ratio of high density lipoprotein/low density lipoprotein levels is substantially increased. Given the inverse relationship between high density lipoprotein levels and coronary heart disease risk, this effect of estrogens on the plasma lipoproteins could be expected to further reduce coronary heart disease risk in women.

Although the bulk of currently available evidence suggests benefit, some controversy concerning the effects of postmenopausal estrogens on morbidity and mortality from coronary heart disease persists. Analysis of the Lipid Research Clinics Follow-up Study population indicated a potentially profound beneficial effect of postmenopausal estrogen use. Mortality from all causes decreased considerably in postmenopausal estrogen users, and the effect was most pronounced in hysterectomized and oophorectomized women. Similar results have been observed for cardiovascular deaths. These benefits appeared to be mediated by the higher high density lipoprotein levels associated with postmenopausal estrogen use. Framingham data are the primary sources reporting possible detrimental effects of postmenopausal estrogen use on cardiovascular morbidity; mortality from all cause and cardiovascular disease was not reported to vary by use.

NHLBI convened a Trans-NIH Estrogen Working Group to make recommendations to NHLBI on the feasibility of undertaking a clinical trial of the effects of postmenopausal estrogen use on cardiovascular disease mortality. The Working Group identified a number of important research questions which needed to be answered to elucidate the effects of postmenopausal estrogen use on risk factors for cardiovascular disease and osteoporosis. This initiative was the result of the Working Group's deliberations and recommendations.

DESIGN NARRATIVE:

There were seven clinical centers and a coordinating center in this randomized, double-blind clinical trial. The women were allocated to one of five treatment arms: placebo; conjugated equine estrogen (CEE), 0.625 milligrams per day; conjugated equine estrogen, 0.625 milligrams per day plus cyclic medroxyprogesterone acetate (MPA), 10 milligrams per day for 12 days per month; CEE, 0.625 milligrams per day plus consecutive MPA, 2.5 milligrams per day; CEE, 0.625 milligrams per day plus cyclic micronized progesterone (MP), 200 milligrams per day for 12 days a month. The four primary endpoints were chosen to represent four biological systems related to the risk of cardiovascular disease and included high density lipoprotein cholesterol (HDL-C), systolic blood pressure, serum insulin, and fibrinogen. Recruitment began in October 1989 and ended in February 1991. Baseline data collected included blood pressure, resting heart rate, weight, waist/hip ratios and endometrial biopsy. Laboratory evaluations included lipid panel, high density lipoprotein cholesterol, insulin and glucose, bone density, fibrinogen, and in three clinics, additional hemostasis factors, renin substrate, plasma renin activity, aldosterone, and oral post-heparin lipase activity. All women underwent an endometrial aspiration biopsy at baseline and annually thereafter. Additional biopsy specimens were obtained if there was noncyclic endometrial bleeding. All women also had baseline and annual mammograms. Other data were collected on quality of life, exercise, diet, alcohol use, and smoking. Participants were followed at three, six and twelve months post-randomization, and at six month intervals thereafter for three years. Post-trial analyses of existing data sets were funded for three years by the cooperative agreement mechanism beginning August 1, 1994. A three-year safety follow-up funded through the contract mechanism began in 1994. It included three annual visits at which endometrial biopsies, mammograms, and some limited health information were obtained.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Postmenopausal women, ages 45 to 64. One third of the subjects had had a hysterectomy.

Ages: 45 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1987-09; Study Completion 2000-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Espeland — Bowman Gray School of Medicine

REFERENCES:
- [Background] Effects of hormone therapy on bone mineral density: results from the postmenopausal estrogen/progestin interventions (PEPI) trial. The Writing Group for the PEPI. JAMA. 1996 Nov 6;276(17):1389-96. PMID 8892713
- [Background] Effects of estrogen or estrogen/progestin regimens on heart disease risk factors in postmenopausal women. The Postmenopausal Estrogen/Progestin Interventions (PEPI) Trial. The Writing Group for the PEPI Trial. JAMA. 1995 Jan 18;273(3):199-208. PMID 7807658
- [Background] Healy B. PEPI in perspective. Good answers spawn pressing questions. JAMA. 1995 Jan 18;273(3):240-1. doi: 10.1001/jama.273.3.240. No abstract available. PMID 7807665
- [Background] National Heart , Lung and Blood Institute. Hormone replacement therapy and heart disease: The PEPI trial. DHHS. NIH Publication No.95-3277. August 1995
- [Background] Effects of hormone replacement therapy on endometrial histology in postmenopausal women. The Postmenopausal Estrogen/Progestin Interventions (PEPI) Trial. The Writing Group for the PEPI Trial. JAMA. 1996 Feb 7;275(5):370-5. doi: 10.1001/jama.1996.03530290040035. PMID 8569016
- [Background] Bush TL, Espeland MA, Mebane-Sims I. The Postmenopausal Estrogen/Progestin Interventions (PEPI) Trial. Introduction. Control Clin Trials. 1995 Aug;16(4 Suppl):1S-2S. doi: 10.1016/0197-2456(94)00119-n. No abstract available. PMID 7587216
- [Background] Espeland MA, Bush TL, Mebane-Sims I, Stefanick ML, Johnson S, Sherwin R, Waclawiw M. Rationale, design, and conduct of the PEPI Trial. Postmenopausal Estrogen/Progestin Interventions. Control Clin Trials. 1995 Aug;16(4 Suppl):3S-19S. doi: 10.1016/0197-2456(95)91154-3. PMID 7587218
- [Background] Johnson S, Mebane-Sims I, Hogan PE, Stoy DB. Recruitment of postmenopausal women in the PEPI Trial. Postmenopausal Estrogen/Progestin Interventions. Control Clin Trials. 1995 Aug;16(4 Suppl):20S-35S. doi: 10.1016/0197-2456(94)00111-f. No abstract available. PMID 7587217
- [Background] Wood PD, Kessler G, Lippel K, Stefanick ML, Wasilauskas CH, Wells HB. Physical and laboratory measurements in the PEPI Trial Postmenopausal Estrogen/Progestin Interventions. Control Clin Trials. 1995 Aug;16(4 Suppl):36S-53S. doi: 10.1016/0197-2456(95)96882-c. No abstract available. PMID 7587219
- [Background] Miller VT, Byington RL, Espeland MA, Langer R, Marcus R, Shumaker S, Stern MP. Baseline characteristics of the PEPI participants. Postmenopausal Estrogen/Progestin Interventions. Control Clin Trials. 1995 Aug;16(4 Suppl):54S-65S. doi: 10.1016/0197-2456(94)00113-h. No abstract available. PMID 7587220
- [Background] Stefanick ML, Legault C, Tracy RP, Howard G, Kessler CM, Lucas DL, Bush TL. Distribution and correlates of plasma fibrinogen in middle-aged women. Initial findings of the Postmenopausal Estrogen/Progestin Interventions (PEPI) study. Arterioscler Thromb Vasc Biol. 1995 Dec;15(12):2085-93. doi: 10.1161/01.atv.15.12.2085. PMID 7489228
- [Background] Marcus R, Greendale G, Blunt BA, Bush TL, Sherman S, Sherwin R, Wahner H, Wells B. Correlates of bone mineral density in the postmenopausal estrogen/progestin interventions trial. J Bone Miner Res. 1994 Sep;9(9):1467-76. doi: 10.1002/jbmr.5650090920. PMID 7817832
- [Background] Greendale GA, Bodin-Dunn L, Ingles S, Haile R, Barrett-Connor E. Leisure, home, and occupational physical activity and cardiovascular risk factors in postmenopausal women. The Postmenopausal Estrogens/Progestins Intervention (PEPI) Study. Arch Intern Med. 1996 Feb 26;156(4):418-24. PMID 8607727
- [Background] Barrett-Connor E, Schrott HG, Greendale G, Kritz-Silverstein D, Espeland MA, Stern MP, Bush T, Perlman JA. Factors associated with glucose and insulin levels in healthy postmenopausal women. Diabetes Care. 1996 Apr;19(4):333-40. doi: 10.2337/diacare.19.4.333. PMID 8729156
- [Background] Greendale GA, James MK, Espeland MA, Barrett-Connor E. Can we measure prior postmenopausal estrogen/progestin use? The Postmenopausal Estrogen/Progestin Interventions Trial. The PEPI Investigators. Am J Epidemiol. 1997 Nov 1;146(9):763-70. doi: 10.1093/oxfordjournals.aje.a009352. PMID 9366624
- [Background] Langer RD, Pierce JJ, O'Hanlan KA, Johnson SR, Espeland MA, Trabal JF, Barnabei VM, Merino MJ, Scully RE. Transvaginal ultrasonography compared with endometrial biopsy for the detection of endometrial disease. Postmenopausal Estrogen/Progestin Interventions Trial. N Engl J Med. 1997 Dec 18;337(25):1792-8. doi: 10.1056/NEJM199712183372502. PMID 9400035
- [Background] Barrett-Connor E, Slone S, Greendale G, Kritz-Silverstein D, Espeland M, Johnson SR, Waclawiw M, Fineberg SE. The Postmenopausal Estrogen/Progestin Interventions Study: primary outcomes in adherent women. Maturitas. 1997 Jul;27(3):261-74. doi: 10.1016/s0378-5122(97)00041-8. PMID 9288699
- [Background] Smith EM, Johnson SR, Figuerres EJ, Mendoza M, Fedderson D, Haugen TH, Turek LP. The frequency of human papillomavirus detection in postmenopausal women on hormone replacement therapy. Gynecol Oncol. 1997 Jun;65(3):441-6. doi: 10.1006/gyno.1997.4703. PMID 9190973
- [Background] Espeland MA, Stefanick ML, Kritz-Silverstein D, Fineberg SE, Waclawiw MA, James MK, Greendale GA. Effect of postmenopausal hormone therapy on body weight and waist and hip girths. Postmenopausal Estrogen-Progestin Interventions Study Investigators. J Clin Endocrinol Metab. 1997 May;82(5):1549-56. doi: 10.1210/jcem.82.5.3925. PMID 9141548
- [Background] Espeland MA, Marcovina SM, Miller V, Wood PD, Wasilauskas C, Sherwin R, Schrott H, Bush TL. Effect of postmenopausal hormone therapy on lipoprotein(a) concentration. PEPI Investigators. Postmenopausal Estrogen/Progestin Interventions. Circulation. 1998 Mar 17;97(10):979-86. doi: 10.1161/01.cir.97.10.979. PMID 9529266
- [Background] Legault C, Espeland MA, Wasilauskas CH, Bush TL, Trabal J, Judd HL, Johnson SR, Greendale GA. Agreement in assessing endometrial pathology: the Postmenopausal Estrogen/Progestin Interventions (PEPI) Trial. J Womens Health. 1998 May;7(4):435-42. doi: 10.1089/jwh.1998.7.435. PMID 9611701
- [Background] Greendale GA, Reboussin BA, Sie A, Singh HR, Olson LK, Gatewood O, Bassett LW, Wasilauskas C, Bush T, Barrett-Connor E. Effects of estrogen and estrogen-progestin on mammographic parenchymal density. Postmenopausal Estrogen/Progestin Interventions (PEPI) Investigators. Ann Intern Med. 1999 Feb 16;130(4 Pt 1):262-9. doi: 10.7326/0003-4819-130-4_part_1-199902160-00003. PMID 10068383
- [Background] Espeland MA, Hogan PE, Fineberg SE, Howard G, Schrott H, Waclawiw MA, Bush TL. Effect of postmenopausal hormone therapy on glucose and insulin concentrations. PEPI Investigators. Postmenopausal Estrogen/Progestin Interventions. Diabetes Care. 1998 Oct;21(10):1589-95. doi: 10.2337/diacare.21.10.1589. PMID 9773716
- [Background] Hall SL, Greendale GA. The relation of dietary vitamin C intake to bone mineral density: results from the PEPI study. Calcif Tissue Int. 1998 Sep;63(3):183-9. doi: 10.1007/s002239900512. PMID 9701620
- [Background] Greendale GA, Reboussin BA, Hogan P, Barnabei VM, Shumaker S, Johnson S, Barrett-Connor E. Symptom relief and side effects of postmenopausal hormones: results from the Postmenopausal Estrogen/Progestin Interventions Trial. Obstet Gynecol. 1998 Dec;92(6):982-8. doi: 10.1016/s0029-7844(98)00305-6. PMID 9840563
- [Background] Cushman M, Legault C, Barrett-Connor E, Stefanick ML, Kessler C, Judd HL, Sakkinen PA, Tracy RP. Effect of postmenopausal hormones on inflammation-sensitive proteins: the Postmenopausal Estrogen/Progestin Interventions (PEPI) Study. Circulation. 1999 Aug 17;100(7):717-22. doi: 10.1161/01.cir.100.7.717. PMID 10449693
- [Background] Marcus R, Holloway L, Wells B, Greendale G, James MK, Wasilauskas C, Kelaghan J. The relationship of biochemical markers of bone turnover to bone density changes in postmenopausal women: results from the Postmenopausal Estrogen/Progestin Interventions (PEPI) trial. J Bone Miner Res. 1999 Sep;14(9):1583-95. doi: 10.1359/jbmr.1999.14.9.1583. PMID 10469288
- [Background] Whiteman MK, Cui Y, Flaws JA, Espeland M, Bush TL. Low fibrinogen level: A predisposing factor for venous thromboembolic events with hormone replacement therapy. Am J Hematol. 1999 Aug;61(4):271-3. doi: 10.1002/(sici)1096-8652(199908)61:43.0.co;2-0. PMID 10440916
- [Background] Barnabei VM, Phillips TM, Hsia J. Plasma homocysteine in women taking hormone replacement therapy: the Postmenopausal Estrogen/Progestin Interventions (PEPI) Trial. J Womens Health Gend Based Med. 1999 Nov;8(9):1167-72. doi: 10.1089/jwh.1.1999.8.1167. PMID 10595329
- [Background] Legault C, Stefanick ML, Miller VT, Marcovina SM, Schrott HG. Effect of hormone replacement therapy on the validity of the Friedewald equation in postmenopausal women: the postmenopausal estrogen/progestins interventions (PEPI) trial. J Clin Epidemiol. 1999 Dec;52(12):1187-95. doi: 10.1016/s0895-4356(99)00107-9. PMID 10580781
- [Background] Greendale GA, Espeland M, Slone S, Marcus R, Barrett-Connor E; PEPI Safety Follow-Up Study (PSFS) Investigators. Bone mass response to discontinuation of long-term hormone replacement therapy: results from the Postmenopausal Estrogen/Progestin Interventions (PEPI) Safety Follow-up Study. Arch Intern Med. 2002 Mar 25;162(6):665-72. doi: 10.1001/archinte.162.6.665. PMID 11911720
- [Background] Simon JA, Symons JP. Bleeding patterns of the hormone replacement therapies in the postmenopausal estrogen and progestin interventions trial. Obstet Gynecol. 2003 May;101(5 Pt 1):1020; author reply 1020-1. doi: 10.1016/s0029-7844(03)00113-3. No abstract available. PMID 12738166
- [Background] Lindenfeld EA, Langer RD. Bleeding patterns of the hormone replacement therapies in the postmenopausal estrogen and progestin interventions trial. Obstet Gynecol. 2002 Nov;100(5 Pt 1):853-63. doi: 10.1016/s0029-7844(02)02245-7. PMID 12423841
- [Background] Hu P, Greendale GA, Palla SL, Reboussin BA, Herrington DM, Barrett-Connor E, Reuben DB. The effects of hormone therapy on the markers of inflammation and endothelial function and plasma matrix metalloproteinase-9 level in postmenopausal women: the postmenopausal estrogen progestin intervention (PEPI) trial. Atherosclerosis. 2006 Apr;185(2):347-52. doi: 10.1016/j.atherosclerosis.2005.06.011. Epub 2005 Jul 14. PMID 16023653
- [Background] Abrams FR. The Postmenopausal Estrogen/Progestin Interventions Trial. JAMA. 1995 Dec 6;274(21):1675; author reply 1676. doi: 10.1001/jama.274.21.1675b. No abstract available. PMID 7474268
- [Background] Garg A. The Postmenopausal Estrogen/Progestin Interventions Trial. JAMA. 1995 Dec 6;274(21):1675-6. doi: 10.1001/jama.1995.03530210029022. No abstract available. PMID 7474269